CLINICAL TRIAL: NCT01327105
Title: Use of Transvaginal Ultrasound to Confirm Essure® Micro-insert Placement in Women: Demonstration of Effectiveness
Brief Title: Essure Transvaginal Ultrasound (TVU) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16974; ESS-TVU (Other: Company internal)
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Contraceptive Usage
MeSH Terms: conditions — Contraception Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TVU (Experimental)
  Interventions: Device: TVU

INTERVENTIONS:
Device: TVU — Use of transvaginal ultrasound to determine location of micro-insert

SUMMARY:
The Essure procedure, FDA approved since 2002 and CE Mark approved since 2001, is the first permanent birth control method that can be performed in the comfort of a physician's office without hormones, cutting, burning or the risks associated with general anesthesia or tubal ligation. Soft, flexible inserts are placed in a woman's fallopian tubes through the cervix without incisions. Over the next three months, the body forms a natural barrier around the micro-inserts to prevent sperm from reaching the egg. Three months after the Essure procedure, a doctor performs an Essure Confirmation Test. In the United States, this test is called a hysterosalpingogram and evaluates the location of the inserts and whether the fallopian tubes are blocked. Outside of the United States, a standard x-ray is performed to evaluate the location of the inserts.

The purpose of this study is to evaluate whether a transvaginal ultrasound is an effective method of confirming micro-insert location.

DETAILED DESCRIPTION:
This study has previously been posted by Conceptus, Inc. (USA).

After acquiring Conceptus, Inc., Bayer HealthCare AG (Germany) is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 21 to 44 years of age
* Women who are between 90-300 pounds (40-136 kilograms)
* Women who are scheduled to undergo an Essure micro-insert placement procedure for permanent birth control
* Women who are willing to accept the risk of pregnancy occurring while relying on the Essure device for prevention of pregnancy
* Women who are believed to have two viable fallopian tubes
* Women who are able and willing to provide written informed consent
* Women who have the mental capacity to understand the Informed Consent, comply with the protocol requirements, and provide reliable feedback regarding device wearing
* Women who can be available for all study visits
* Women who are willing to allow data to be shared with the sponsor and with regulatory bodies
* Women who are not contraindicated for the Essure procedure according to the Essure Instructions for Use (IFU)

Exclusion Criteria:

* Women who have known proximal tubal occlusion in either fallopian tube
* Women who have had a fallopian tube sterilization procedure
* Women who have a unicornuate uterus
* Women who have known endometrial or myometrial pathology that is likely to prevent access to the fallopian tube ostia
* Women who are scheduled to undergo any other intrauterine procedures at the time of Essure placement
* Women who are pregnant or suspected of being pregnant
* Women who have had a delivery or termination of pregnancy within the last six weeks
* Women who have an active or recent upper or lower pelvic infection
* Women who are contraindicated for Essure micro-insert placement according to the Essure Instructions for Use (IFU)
* Women who have a known intolerance to transvaginal imaging

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 547 (Actual)
Dates: Start 2011-05-17 (Actual); Primary Completion 2014-07-16 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
Effectiveness | Annually beginning at one year
  Rate of pregnancy at 1 and 10 years among subjects relying on Essure micro-inserts for birth control on the basis of the TVU/HSG algorithm

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (21):
- United States (13):
  - Chandler, Arizona
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Arvada, Colorado
  - Fort Wayne, Indiana
  - Saginaw, Michigan
  - Rochester, Minnesota
  - The Bronx, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Houston, Texas
- Regina, Saskatchewan, Canada
- Netherlands (6):
  - Amsterdam
  - Hoofddorp
  - Nieuwegein
  - Tiel
  - Veldhoven
  - Zwolle
- Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Vleugels M, Cheng RF, Goldstein J, Bangerter K, Connor V. Algorithm of Transvaginal Ultrasound and/or Hysterosalpingogram for Confirmation Testing at 3 Months after Essure Placement. J Minim Invasive Gynecol. 2017 Nov-Dec;24(7):1128-1135. doi: 10.1016/j.jmig.2017.06.021. Epub 2017 Jun 29. PMID 28669895